CLINICAL TRIAL: NCT04836858
Title: A Randomized, Subject and Investigator Blinded, Placebo-controlled Multicenter Study to Assess the Efficacy and Safety of CMK389 in Patients With Moderate to Severe Atopic Dermatitis
Brief Title: A Study to Assess the Efficacy and Safety of CMK389 in Patients With Moderate to Severe Atopic Dermatitis.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CCMK389B12201; 2020-003406-31 (EudraCT Number)
Record Dates: First submitted 2021-03-24; First posted 2021-04-08 (Actual); Results first posted 2024-05-09 (Actual); Last update posted 2024-06-20 (Actual); Status verified 2024-06

CONDITIONS: Atopic Dermatitis
Keywords: Atopic Dermatitis; Safety; Efficacy; Atopic Eczema; Eczema; CMK389
MeSH Terms: conditions — Dermatitis, Atopic; Eczema

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- CMK389 10mg/kg i.v. (Experimental): Active
  Interventions: Biological: CMK389
- Placebo i.v. (Placebo Comparator): Placebo
  Interventions: Biological: Placebo
- CMK389 300mg s.c. (Experimental): Active
  Interventions: Biological: CMK389
- Placebo s.c. (Placebo Comparator): Placebo
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: CMK389 — Active
  Arms: CMK389 10mg/kg i.v.; CMK389 300mg s.c.
Biological: Placebo — Placebo Comparator
  Arms: Placebo i.v.; Placebo s.c.

SUMMARY:
The main purpose of this phase 2 study was to assess the efficacy and safety of CMK389 in patients with atopic dermatitis.

DETAILED DESCRIPTION:
This was a randomized, placebo-controlled, parallel-group, non-confirmatory, investigator and participant blinded study in adult participants with moderate to severe AD. The study consisted of up to 4 weeks screening period to assess participants eligibility, the baseline visit, 4-weekly administrations of CMK389 within the first 12 weeks of the 16-week treatment period, and an approximately 12 weeks follow up period which finished with the end of study visit (EoS). In addition, for women of child-bearing potential, pregnancy tests were done for 6 months after the last dose of CMK389.

ELIGIBILITY:
Inclusion Criteria:

* Adult male or female participants with chronic atopic dermatitis, aged 18 to 65 years, present for at least 1 year before screening.
* Participants with Moderate to severe AD defined by IGA score of ≥ 3 (on a scale of 0 to 4, in which 3 is moderate and 4 is severe) at Baseline, EASI score of ≥ 12 at Baseline and Pruritus (NRS) of at least ≥ 3 at Baseline
* Participants who are candidates for a systemic therapy, defined as e.g. inadequate response to treatment with topical medications, or for whom topical treatments are otherwise medically inadvisable (e.g. because of important side effects or safety risks, patients with large affected body surface areas) as assessed by the investigator.
* Participants must have a body mass index (BMI) at screening within the range of 18 to ≤35 kg/m2.

Exclusion Criteria:

* Any skin disease that, in the opinion of the investigator, would confound the diagnosis or evaluation of AD disease activity.
* Participants taking prohibited medication not completing the wash out period
* Use of other investigational drugs at the time of enrolment, or within 5 half-lives of enrolment, or until the expected PD effect has returned to baseline, whichever is longer; or longer if required by local regulations.
* Any active, recent or recurrent systemic or localized infection at screening or prior to first treatment which in the opinion of the investigator immunocompromises the participant and/or places the participant at unacceptable risk for immunomodulatory therapy, such as:

  * Any acute bacterial, fungal, or viral skin/mucosal infection that has not resolved within 2 weeks prior to first treatment or within 12 months in case of eczema herpeticum.
  * Clinically infected AD within 4 weeks prior to first treatment.
  * Any other infection requiring treatment with systemic antibiotics, antivirals, antiparasitics, antiprotozoals, or antifungals within 4 weeks prior to first treatment.
  * Tuberculosis (TB), Human Immunodeficiency Virus (HIV), Hepatitis B, Hepatitis C
* Any other current or past clinically significant medical condition, including psychiatric condition, which in the Investigator's opinion may interfere with safety of the participant, study objectives or adherence to the protocol.
* Participants with confirmed abnormal absolute neutrophil count (ANC) of <1.5 x 10^9/L or with thrombocytopenia of < 75.0 x 10^9/L at screening and baseline
* History of malignancy of any organ system (other than localized basal cell carcinoma of the skin), treated or untreated, within the past 5 years, regardless of whether there is evidence of local recurrence or metastases.
* History of hypersensitivity to any component of the study drug product, or to drugs of similar chemical classes.
* History of severe or serious allergy or hypersensitivity reactions, such as anaphylactic shock, asthma, or uncontrolled urticaria.
* Pregnant or nursing (lactating) women.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2021-04-20 (Actual); Primary Completion 2022-07-14 (Actual); Study Completion 2022-12-13 (Actual)

CONTACTS AND LOCATIONS:
Locations (18):
- Czechia (2):
  - Novartis Investigative Site, Pardubice, Czech Republic
  - Novartis Investigative Site, Prague
- France (3):
  - Novartis Investigative Site, Marseille
  - Novartis Investigative Site, Nice
  - Novartis Investigative Site, Rouen
- Germany (7):
  - Novartis Investigative Site, Bad Bentheim
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Frankfurt
  - Novartis Investigative Site, Heidelberg
  - Novartis Investigative Site, München
  - Novartis Investigative Site, Münster
  - Novartis Investigative Site, Osnabrück
- Hungary (2):
  - Novartis Investigative Site, Budapest
  - Novartis Investigative Site, Szeged
- Poland (3):
  - Novartis Investigative Site, Gdansk
  - Novartis Investigative Site, Lodz
  - Novartis Investigative Site, Rzeszów
- Novartis Investigative Site, Córdoba, Andalusia, Spain

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- See also: Patient Lay Trial Summary — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=1800

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in 18 investigative sites in 6 countries.
Pre-assignment Details: There was a screening period of up to 4 weeks to assess participants eligibility.
Groups:
- CMK389 10mg/kg i.v.: CMK389 10 mg/kg monthly i.v. dose
- CMK389 300mg s.c.: CMK389 300mg monthly s.c. dose
- Placebo i.v.: Placebo monthly i.v. dose
- Placebo s.c.: Placebo monthly s.c. dose
Period: Overall Study
Arm/Group | CMK389 10mg/kg i.v. | CMK389 300mg s.c. | Placebo i.v. | Placebo s.c.
Started (All participants randomized in the trial.) | 38 | 17 | 8 | 8
Safety Analysis Set (All participants who received any study drug.) | 34 | 17 | 8 | 8
Completed | 30 | 17 | 8 | 6
Not Completed | 8 | 0 | 0 | 2
Not completed — Adverse Event | 0 | 0 | 0 | 1
Not completed — Lost to Follow-up | 1 | 0 | 0 | 0
Not completed — Subject/Guardian decision | 3 | 0 | 0 | 1
Not completed — Randomized but not treated | 4 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety analysis set defined as all participants who received any study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | CMK389 10mg/kg i.v. | CMK389 300mg s.c. | Placebo i.v. | Placebo s.c. | Total
Number analyzed (Participants) | 34 | 17 | 8 | 8 | 67
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.7 (9.86) | 34.1 (11.35) | 35.3 (8.86) | 31.9 (8.53) | 33.8 (9.83)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 9 | 3 | 2 | 22
  Male | 26 | 8 | 5 | 6 | 45
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 0 | 1 | 0 | 0 | 1
  White | 34 | 16 | 8 | 8 | 66

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Investigator Global Assessment (IGA) Response
Description: The Investigator Global assessment (IGA) scale used was vIGA-AD^TM (Validated Investigator Global Assessment scale for Atopic Dermatitis). The IGA rating scale was used to determine the severity of atopic dermatitis and clinical response to treatment. It reflected a participant's overall disease severity for the whole body based on a 5-point scale. The 5-point scale included: clear, almost clear, mild, moderate, and severe disease. IGA response is defined as clear or almost clear and at least a 2 point-reduction from baseline at week 16.
Time Frame: Baseline, Week 16
Population: The safety analysis set included all participants who received any study drug.
Measure: Count of Participants; unit: Participants
Groups:
- Pooled Placebo: Pooled Placebo monthly i.v. and s.c. dose
Arm/Group | CMK389 10mg/kg i.v. | CMK389 300mg s.c. | Placebo i.v. | Placebo s.c. | Pooled Placebo
Number analyzed (Participants) | 34 | 17 | 8 | 8 | 16
Participants | 5 | 2 | 0 | 0 | 0

2. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: Number of participants with treatment emergent AEs (any AE regardless of seriousness), AEs led to study treatment discontinuation, SAEs and SAEs led to study treatment discontinuation.
Time Frame: AEs were reported from first dose until the end of the 12 weeks follow up period, up to a max. duration of approx. 197 days. For women of child-bearing potential, pregnancies were reported (if occurred) for up to approx. 268 days after first dose.
Population: The safety analysis set included all participants who received any study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | CMK389 10mg/kg i.v. | CMK389 300mg s.c. | Placebo i.v. | Placebo s.c.
Number analyzed (Participants) | 34 | 17 | 8 | 8
Participants
  Adverse Events | 25 | 11 | 5 | 8
  Serious Adverse Events | 1 | 1 | 0 | 0
  AEs leading to discontinuation of study treatment | 0 | 0 | 0 | 0
  SAEs leading to discontinuation of study treatment | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: AEs were reported from first dose until the end of the 12 weeks follow up period, up to a max. duration of approx. 197 days. For women of child-bearing potential, pregnancies were reported (if occurred) for up to approx. 268 days after first dose.
Groups:
- CMK389 10 mg/kg i.v.: CMK389 10 mg/kg monthly i.v. dose
- CMK389 300 mg s.c.: CMK389 300mg monthly s.c. dose
- Total: Total
Arm/Group | CMK389 10 mg/kg i.v. | CMK389 300 mg s.c. | Placebo i.v. | Placebo s.c. | Pooled Placebo | Total
All-Cause Mortality (participants affected / at risk) | 0/34 | 0/17 | 0/8 | 0/8 | 0/16 | 0/67
Serious Adverse Events (participants affected / at risk) | 1/34 | 1/17 | 0/8 | 0/8 | 0/16 | 2/67
Other Adverse Events (participants affected / at risk) | 20/34 | 11/17 | 5/8 | 8/8 | 13/16 | 44/67
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CMK389 10 mg/kg i.v. (N=34) | CMK389 300 mg s.c. (N=17) | Placebo i.v. (N=8) | Placebo s.c. (N=8) | Pooled Placebo (N=16) | Total (N=67)
Heavy menstrual bleeding (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 1
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | CMK389 10 mg/kg i.v. (N=34) | CMK389 300 mg s.c. (N=17) | Placebo i.v. (N=8) | Placebo s.c. (N=8) | Pooled Placebo (N=16) | Total (N=67)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 1
Sinus bradycardia (Cardiac disorders) | 0 | 0 | 1 | 0 | 1 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0 | 1
Eyelid oedema (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 1
Visual impairment (Eye disorders) | 0 | 1 | 1 | 0 | 1 | 2
Diarrhoea (Gastrointestinal disorders) | 3 | 2 | 0 | 0 | 0 | 5
Nausea (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 1
Fatigue (General disorders) | 0 | 0 | 1 | 0 | 1 | 1
Injection site reaction (General disorders) | 0 | 1 | 0 | 0 | 0 | 1
Asymptomatic bacteriuria (Infections and infestations) | 0 | 0 | 0 | 1 | 1 | 1
Bacteriuria (Infections and infestations) | 0 | 0 | 1 | 0 | 1 | 1
COVID-19 (Infections and infestations) | 10 | 5 | 3 | 1 | 4 | 19
Nasopharyngitis (Infections and infestations) | 7 | 4 | 1 | 1 | 2 | 13
Otitis externa (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 1
Rhinitis (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 2
Upper respiratory tract infection (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 2
Alanine aminotransferase increased (Investigations) | 2 | 0 | 0 | 0 | 0 | 2
Aspartate aminotransferase increased (Investigations) | 2 | 0 | 0 | 0 | 0 | 2
Blood creatine increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 1
Blood creatine phosphokinase increased (Investigations) | 2 | 0 | 0 | 1 | 1 | 3
Blood ketone body increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 1
Glucose urine (Investigations) | 0 | 1 | 0 | 0 | 0 | 1
Lymphocyte count decreased (Investigations) | 0 | 0 | 0 | 1 | 1 | 1
Urinary sediment present (Investigations) | 0 | 0 | 1 | 0 | 1 | 1
Urine analysis abnormal (Investigations) | 0 | 0 | 1 | 0 | 1 | 1
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 1 | 1
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0 | 0 | 2
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 1 | 1
Muscle tightness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 1 | 1
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 3 | 1 | 1 | 0 | 1 | 5
Migraine (Nervous system disorders) | 0 | 0 | 2 | 0 | 2 | 2
Hypertonic bladder (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 1
Menstruation irregular (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 1
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 1 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 1
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 1 | 1
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 2 | 2 | 0 | 4 | 4 | 8
Psoriasis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 1
Hypertension (Vascular disorders) | 0 | 2 | 0 | 0 | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2022-03-04): https://cdn.clinicaltrials.gov/large-docs/58/NCT04836858/Prot_000.pdf
  • Statistical Analysis Plan (2023-01-12): https://cdn.clinicaltrials.gov/large-docs/58/NCT04836858/SAP_001.pdf